CLINICAL TRIAL: NCT01820403
Title: Portion Size Effects on Body Weight: Free Living Setting
Brief Title: Portion Size Effects on Body Weight:Free Living Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FWA00000312-3; R01DK081714 (NIH)
Record Dates: First submitted 2013-03-25; First posted 2013-03-28 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Portion Sizes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- portion size small (Experimental): 400 kcal box lunch was delivered each weekday to each participant at the worksite for a six month period.
  Interventions: Other: portion size kcal of box lunch
- portion size medium (Experimental): 800 kcal box lunch was delivered each weekday to each participant at the worksite for a six month period.
  Interventions: Other: portion size kcal of box lunch
- portion size large (Experimental): 1600 kcal box lunch was delivered each weekday to each participant at the worksite for a six month period.
  Interventions: Other: portion size kcal of box lunch
- control (No Intervention): no box lunch provided to participants.

INTERVENTIONS:
Other: portion size kcal of box lunch
  Other Names: box lunches of different portion sizes were provided to participants each weekday for six months. Portion size conditions were 440 kcal, 800 kcal or 1600 kcal.
  Arms: portion size large; portion size medium; portion size small

SUMMARY:
The study purpose was to evaluate the effects of portion sizes on body weight and energy intake in a free-living setting. 223 healthy adults were recruited from an urban worksite and randomized to one of four groups for a six-month period. The groups were: 1) 400 kcal box lunch; 2) 800 kcal box lunch; 3) 1600 kcal box lunch; or 4) no box lunch. Participants were required to pick up a box lunch every week day for six months. Control participants did not receive a box lunch and were instructed to eat their usual lunch. Participants were weighed and dietary intake measured at baseline, one, three and six months. It was hypothesized that at six months, participants in the 1600 kcal box lunch would gain more weight and have higher energy intake than those in the other groups.

ELIGIBILITY:
Inclusion Criteria:

* : 1) age 18-60 yrs; 2) nonsmoker; 3) fluent in English; 4) not taking medications that affect appetite or body weight; 5) work at the medical complex full time, including during the lunch hours; 6) not allergic to the foods in the study lunches; 7) willing to eat the foods in the study lunches [examples were provided of the types of foods]; 8) not currently on a diet to lose weight; 9) no history of a diagnosed eating disorder; 10) not moving from the area during the next six months; 11) not currently taking part in another research study; 12) not currently pregnant, nursing or pregnant in the last 12 months.

Exclusion Criteria: if the person does not meet the criteria above

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 233 (Actual)
Dates: Start 2010-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
body weight change | six months
  change in body weight from baseline to six months

SECONDARY OUTCOMES:
dietary energy intake | six months
  change in energy intake from baseline to six months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States